CLINICAL TRIAL: NCT00322062
Title: A Prospective Randomised Single-Blinded Multicentric and Pivotal Phase III Study Comparing the Efficacy, Safety and Acceptability of a New 2 Litres Gut Lavage Solution NRL994 Versus a Sodium Phosphate Solution for Colonoscopy Preparation
Brief Title: MOVIPREP® Versus NaP Pivotal Phase III Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Dr Marc Halphen, Norgine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRL994-02/2001
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Colonoscopy
Keywords: Colon cleansing
MeSH Terms: interventions — MoviPrep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 1 pack (contains 4 (2 x PEG + E/"P" + 2 x Vitamin C/"C") sachets)= 2L NRL994 . 2 sachets (one of each) will be dissolved in 1L of water. Each litre will be drunk within 1 hour. Furthermore, at least 1000ml (or more) of any additional clear fluid (except milk) has to be drunk after the 2L of NRL994.
  Interventions: Drug: macrogol3350 NA sulphate NACL KCL ascorbic acid NA ascorbate
- 2 (Active Comparator): 1 pack consists of 2 flasks of 45ml. Each flask has to be dissolved within 125ml of water. Each intake of NaP solution has to be preceded and followed by 250ml (or more if necessary)of clear liquids(excluding milk)and a delay of at least 12 hours between the intake of the 2 x 45ml of NaP solution has to be completed. In addition, 750ml more of clear liquids (excluding milk)or more if needed must be drunk between the 2 intakes.
  Interventions: Drug: Sodium Phosphate Solution

INTERVENTIONS:
Drug: macrogol3350 NA sulphate NACL KCL ascorbic acid NA ascorbate — 2L gut lavage solution
  Other Names: MOVIPREP®
  Arms: 1
Drug: Sodium Phosphate Solution — 1 x 45ml solution, BID
  Other Names: Fleet Phospho Soda®
  Arms: 2

SUMMARY:
The aim of the study is to compare a new 2 litre bowel cleansing product versus a sodium phosphate solution already on the market. Efficacy of each bowel preparation, safety and acceptability will be assessed.

DETAILED DESCRIPTION:
Multicentric (15 centres), prospective, randomised, single-blinded phase III pivotal study in patients undergoing a colonoscopy. Gut cleansing will be performed using 2 litres of NRL994 gut lavage solution with 1 litre (or more) of extra clear liquids or 2 x 45 ml of a sodium phosphate solution plus 2 litres (or more) of extra clear liquids the day before colonoscopy. Patients requiring a morning colonoscopy who fulfil the inclusion criteria, will be randomised. One of the two tested products will be delivered by a pharmacist, blindly from the gastroenterologist. The assigned product will be taken the day before the coloscopy according to the information leaflet. Efficacy of the two tested preparations will be measured on video-tape record of each colonoscopy by a final grading i.e. "the overall quality of colonoscopy prep" by an gastroenterologist expert. A standardised patient questionnaire administered by a nurse on the morning before colonoscopy will assess clinical tolerance and acceptability (satisfaction) of the prep. A baseline blood sampling will be withdrew before intake of the preparation and one more blood sample will be performed after the intake on the morning, before the coloscopy.

After the coloscopy, as the gastroenterologist gives the result of the coloscopy , a last visit is performed.

ELIGIBILITY:
Inclusion Criteria:

* male or female, out and inpatients to be at least 18 years old and <75 years old sent to the endoscopic ward for diagnostic or therapeutic colonoscopy
* willing and able to complete the entire procedure and to comply with study instructions
* females of childbearing potential must employ an adequate method of contraception.

Exclusion Criteria:

* age <18 or > 75 years old
* ileus
* suspected intestinal occlusion or perforation
* toxic or congenital megacolon
* history of colonic resection
* patients with Crohn's disease or ulcerative colitis
* congestive heart failure NYHA III or IV
* documented renal insufficiency history with creatinine >170µmol/l
* known hypersensitivity to polyethylene glycols or Na phosphate and/or vitamin C
* concurrent participation in an investigational drug study or participation within 90 days of study entry
* females who are pregnant, or planning a pregnancy. Females of childbearing potential not using reliable methods of contraception
* subject has a condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound the study results, or may interfere significantly

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2002-04; Study Completion 2003-03

PRIMARY OUTCOMES:
efficacy will be measured and graded using video-taped record of each colonoscopy for cleansing in a 0 - 4 grade scale for each of the predefined colon areas by an endoscopist.
Grades A or B means a good or correct preparation and are considered as a success whilst C or D are considered as a failed preparation.

SECONDARY OUTCOMES:
evaluation of the preparation quality using a visual analogue scale
recording adverse events and clinical tolerance
patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Alain Bitoun, MD, Principal Investigator — Hôpital Lariboisère
Locations (18):
- France (18):
  - Hôpital Jean Minjoz, Besançon
  - Hôpital Mourier, Colombes
  - Hôpital Huriez, Lille
  - Hôpital Dupuytren, Limoges
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Nord, Marseille Nord Cedex 20
  - Centre Hospitalier, Montélimar
  - Centre Hospitalier Intercommunal, Montfermeil
  - Centre Hospitalier De Montpellier Hôpital St Eloi, Montpellier
  - Hôpital De L'Archet, Nice
  - Hôpital Bichat Claude Bernard, Paris
  - Hôpital Croix Saint Simon, Paris
  - Hôpital Cochin, Paris
  - Unité Endoscopies Digestives, Hôpital Lariboisière, 2 rue Ambroise Paré, Paris
  - Hôpital Civil / Clinique Medical B, Strasbourg
  - Hôpital Rangueil, Toulouse
  - Hôpital Trousseau CHRU, Tours
  - CHU De Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Fordtran JS, Santa Ana CA, Cleveland MvB. A low-sodium solution for gastrointestinal lavage. Gastroenterology. 1990 Jan;98(1):11-6. doi: 10.1016/0016-5085(90)91284-d. PMID 2293568